CLINICAL TRIAL: NCT06177691
Title: Hybrid Closed Loop Therapy and Verapamil for Beta Cell Preservation in New Onset Type 1 Diabetes (CLVer): Extension Study
Acronym: CLVerEx
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CLVerEx
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Type1 Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Participants with body weight ≥30 kg (Cohort A) were randomly assigned in a factorial design during the RCT to (1) HCL plus intensive diabetes management or usual care with no HCL and (2) verapamil or placebo. No interventions were administered during the observational extension.
- Cohort B: Participants with body weight <30 kg (Cohort B) were randomly assigned during the RCT 2:1 in a parallel group design to HCL plus intensive diabetes management or to usual care with no HCL. No interventions were administered during the observational extension.

SUMMARY:
The purpose of this extension study is to continue to follow the participants who completed the CLVer RCT for up to 3 additional years. The goal for Cohort A is to evaluate the longer-term effects of verapamil on preservation of β-cell function as measured by C-peptide levels obtained during a mixed meal tolerance test (MMTT). For both Cohorts A and B, the goal is to determine if the high degree of glycemic control achieved during CLVer with HCL can be maintained once the intensive engagement of the study team is discontinued. At the completion of the RCT, study treatments end. Thus, during the extension study, diabetes management is performed as part of usual care and there is no study treatment.

DETAILED DESCRIPTION:
Participants who complete the CLVer RCT will be eligible to enroll in the CLVer Extension Study. Informed consent and assent, when applicable, will be obtained. Participants will be contacted every 3 months at which time continuous glucose monitoring (CGM) data will be obtained if a CGM device is being used and medical history (including recent point-of-care or local laboratory HbA1c values) will be reviewed; a usual care visit performed by study staff may be considered a study contact. A study visit will occur yearly to update the diabetes and medical history, measure height and weight, determine Tanner staging, download CGM data if available, perform an MMTT, and obtain blood samples for central lab measurement of HbA1c and plasma for storage if consented. Other than the central lab samples, there are no study-specific procedures or data collection that would not be performed as part of standard care.

ELIGIBILITY:
Completed CLVer RCT 12 month visit and willing to join observational extension.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants who complete the CLVer RCT 12 month visit. RCT participants were youth aged 7-<18 years at RCT screening with newly diagnosed stage 3 type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
C-peptide | Randomization, 13, 26, 39 weeks, Year 1, Year 2, Year 3, Year 4
  The primary outcome is the C-peptide measured during the MMTT annually. This is measured as the area under the stimulated C-peptide curve (AUC). AUC is computed using a trapezoidal rule, which is a weighted sum of the C-peptide values over the 120 min. Peak C-peptide also will be computed.

SECONDARY OUTCOMES:
HbA1c | Randomization, 13, 26, 39 weeks, Year 1, Year 2, Year 3, Year 4
  HbA1c outcomes, measured annually, will include the following:
  * Mean HbA1c
  * Percentage of participants with an HbA1c <7.5%, <7.0% and <6.5%
CGM Metrics | 6, 13, 26, 39 weeks, Year 1, Year 2, Year 3, Year 4
  CGM metrics will be computed for each time point of data collection. CGM-derived indices will be computed for 24 hours, daytime (6AM to midnight) and nighttime (midnight to 6AM). The Statistical Analysis Plan (SAP) will describe how CGM derived indices will be calculated. The following metrics will be computed:
  * Mean glucose
  * Percentage of sensor glucose from 70 to 180 mg/dL
  * Percentage of sensor glucose >180 and >250 mg/dL
  * Percentage of sensor glucose <54 and <70 mg/dL
  * Coefficient of variation
Severe hypoglycemia episodes | Year 4
  Frequency of episodes of severe hypoglycemia by cohort group.
Diabetic ketoacidosis events | Year 4
  Frequency of episodes of diabetic ketoacidosis by cohort group.
Hospitalizations | Year 4
  Frequency of hospitalizations by cohort group.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, MD, Study Chair — University of Minnesota; Gregory Forlenza, MD, Study Chair — Barbara Davis Center
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri